CLINICAL TRIAL: NCT02462421
Title: Pharmacogenetics of Sodium-dependent Glucose Transporter-2 (SGLT2) Inhibitors
Brief Title: Pharmacogenetics of SGLT2 Inhibitors
Acronym: SGLT2iPGx
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not meet recruitment targets.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Simeon I. Taylor, Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00058350; R21DK105401 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-06-04 (Estimated); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus; Gout; Hyperuricemia
Keywords: SGLT2; SLC5A2; SLC5A4; SLC5A9; SLC2A9; GLUT9; SGLT3; SGLT4; pharmacogenomics
MeSH Terms: conditions — Diabetes Mellitus; Gout; Hyperuricemia | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Wild type genotype (Active Comparator): Research subjects with wild type genotypes at three candidate genes encoding sodium-dependent glucose transporter-3, sodium-dependent glucose transporter-4, and glucose transporter-9 (abbreviated as SLC5A4, SLC5A9, SLC2A9, respectively) will be studied before and after canagliflozin treatment.
  Interventions: Drug: Canagliflozin
- Nonsense mutation in SLC5A4 (Experimental): Research subjects who are homozygous for nonsense mutation in SLC5A4 (sodium-dependent glucose transporter-3) will be studied before and after canagliflozin treatment.
  Interventions: Drug: Canagliflozin
- Nonsense mutation in SLC5A9 (Experimental): Research subjects who are homozygous for nonsense mutation in SLC5A9 (sodium-dependent glucose transporter-4) will be studied before and after canagliflozin treatment.
  Interventions: Drug: Canagliflozin
- Missense variant in SLC2A9 (Experimental): Research subjects who are homozygous for nonsynonymous variant in glucose transporter-9 (SLC2A9) will be studied before and after canagliflozin treatment.
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — A single dose of canagliflozin (300 mg, p.o.) will be administered prior to assessing pharmacodynamic response.
  Other Names: Invokana

SUMMARY:
Sodium-dependent glucose transporter-2 (SGLT2) inhibitors are a new class of anti-diabetic drugs, which increase urinary glucose excretion thereby promoting weight loss and decreasing plasma glucose levels. We hypothesize that the pharmacodynamic response to SGLT2 inhibitors (specifically canagliflozin) varies among individuals, and that a proportion of this inter-individual variation can be explained by genetic variation. This is a pilot study in healthy, non-diabetic subjects in whom glucose and other related metabolites in the urine and plasma will be measured before and after administration of a single dose of canagliflozin. This will allow us to characterize the inter-individual variation in the pharmacodynamic response to canagliflozin as well as determine if changes in glucose and other related metabolite levels are associated with variants in various candidate genes.

DETAILED DESCRIPTION:
Sodium-dependent glucose transporters (SGLTs) are a family of glucose transporters expressed on the apical surface of epithelial cells in the intestines and kidneys. Their function is to actively transport glucose across epithelia into the blood. Members of the SGLT-family of transporters include sodium-dependent glucose transporters-1, -2, -3, and -4 (SGLT1, SGLT2, SGLT3 and SGLT4), with SGLT2 being the primary glucose transporter in the kidney. SGLT2 inhibitors are a new class of anti-diabetic drug approved as treatments for type 2 diabetes (T2DM). These drugs inhibit SGLT2-mediated reabsorption of glucose in the renal proximal tubule -- thereby increasing urinary glucose excretion and decreasing plasma glucose levels. We hypothesize that the pharmacodynamic response to SGLT2 inhibitors (specifically canagliflozin) varies among individuals, and that a proportion of this inter-individual variation can be explained by genetic variation. To explore this hypothesis, we will conduct a pilot study in healthy, non-diabetic subjects in whom glucose and other related metabolites in the urine and plasma will be measured before and after administration of a single dose of canagliflozin. This will allow us to characterize the inter-individual variation in the pharmacodynamic response to canagliflozin as well as determine if changes in glucose and other related metabolite levels are associated with variants in candidate genes (SGLT3, SGLT4, and glucose transporter-2 (abbreviated as either GLUT9 or SLC2A9)).

ELIGIBILITY:
Inclusion Criteria:

* Of Amish descent
* Age 21 or older
* BMI 18-40 kg/m2

Exclusion Criteria:

* Known allergy to canagliflozin
* History of diabetes, random glucose greater than 200 mg/dL, or HbA1c greater than or equal to 6.5%
* Currently taking diuretics, antihypertensive medication, uric acid lowering medications, or other medication that the investigator judges will make interpretation of the results difficult
* Significant debilitating chronic cardiac, hepatic, pulmonary, or renal disease or other diseases that the investigator judges will make interpretation of the results difficult or increase the risk of participation
* Seizure disorder
* Positive urine human chorionic gonadotropin (hCG) test or known pregnancy within 3 months of the start of the study
* Estimated glomerular filtration rate less than 60 mL/min
* Currently breast feeding or breast feeding within 3 month of the start of the study
* Liver function tests greater than 2 times the upper limit of normal
* Hematocrit less than 35%
* Currently symptomatic for urinary tract or yeast infection or history of two or more urinary tract or yeast infections in the past 12 months.
* Abnormal thyroid stimulating hormone (TSH)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simeon I Taylor, MD, PhD, Study Chair — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in order to protect confidentiality of research subjects.

REFERENCES:
- [Derived] Taylor SI, Montasser ME, Yuen AH, Fan H, Yazdi ZS, Whitlatch HB, Mitchell BD, Shuldiner AR, Muniyappa R, Streeten EA, Beitelshees AL. Acute pharmacodynamic responses to exenatide: Drug-induced increases in insulin secretion and glucose effectiveness. medRxiv [Preprint]. 2023 May 3:2023.03.15.23287166. doi: 10.1101/2023.03.15.23287166. PMID 36993363
- [Derived] Taylor SI, Cherng HR, Yazdi ZS, Montasser ME, Whitlatch HB, Mitchell BD, Shuldiner AR, Streeten EA, Beitelshees AL. Pharmacogenetics of SGLT2 Inhibitors: Validation of a sex-agnostic pharmacodynamic biomarker. medRxiv [Preprint]. 2023 Jun 12:2023.03.07.23286875. doi: 10.1101/2023.03.07.23286875. PMID 36945579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We over-estimated the percentage of people who would agree to participate in this clinical trial. Ultimately, we terminated the study after 30 participants had completed the clinical trial.
Period: Overall Study
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9
Started | 13 | 4 | 6 | 7
Completed | 13 | 4 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
Age, Continuous [Mean (Full Range); unit: Years] | 58.6 [35 to 77] | 57.5 [49 to 70] | 58.2 [37 to 82] | 56.1 [37 to 73] | 57.8 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 4 | 3 | 17
  Male | 4 | 3 | 2 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 4 | 6 | 7 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 13 | 4 | 6 | 7 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 4 | 6 | 7 | 30
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (5.3) | 30.1 (3.5) | 28.2 (5.9) | 25.7 (3.2) | 28.0 (4.8)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.72 (0.15) | 0.79 (0.08) | 0.74 (0.13) | 0.75 (0.11) | 0.74 (0.12)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 95.3 (14.6) | 96.5 (8.3) | 96.0 (14.3) | 98.0 (17.1) | 96.4 (13.9)
Serum sodium [Mean (Standard Deviation); unit: mEq/L] | 138.8 (1.3) | 138.0 (1.8) | 138.7 (1.2) | 137.6 (1.5) | 138.4 (1.4)
HbA1c [Mean (Standard Deviation); unit: % of total hemoglobin that is glycated] | 5.8 (0.2) | 5.7 (0.2) | 5.8 (0.2) | 5.5 (0.4) | 5.7 (0.3)
Hematocrit [Mean (Standard Deviation); unit: %] | 41.8 (2.4) | 43.8 (4.5) | 39.9 (4.3) | 43.3 (3.1) | 42.0 (3.3)
Serum uric acid level [Mean (Standard Deviation); unit: mg/dL] | 4.60 (0.72) | 5.25 (0.55) | 4.05 (1.53) | 3.74 (0.71) | 4.38 (0.93)
creatinine clearance [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 110 (29) | 118 (31) | 103 (18) | 126 (37) | 113 (30)
Fractional excretion of uric acid [Mean (Standard Deviation); unit: % of filtered uric acid that is excreted] | 8.0 (1.3) | 9.4 (3.7) | 6.2 (1.5) | 9.8 (2.9) | 8.5 (2.4)
Urinary sodium excretion (24 hr) [Mean (Standard Deviation); unit: mEq/day] | 196 (50) | 182 (38) | 208 (105) | 247 (68) | 208 (67)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Excretion of Glucose (Measured During the 24 Hours Following Administration of Canagliflozin)
Description: The pharmacodynamic response to canagliflozin will be assessed by measuring the increase in 24 hour urinary glucose excretion.
Time Frame: 24 hours after administration of canagliflozin
Population: The entire population of 30 research participants comprised the database for this analysis.
Measure: Mean (Standard Error); unit: glucose (g)/creatinine (g)
Groups:
- Total Population: Aggregate of all research participants in the four genotypes comprising the four arms of the study.
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total Population
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
glucose (g)/creatinine (g) | 37.6 (2.1) | 37.1 (3.3) | 39.1 (2.5) | 36.9 (2.7) | 37.7 (1.2)
Statistical Analysis 1: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A4; Each of the variant genotypes was compared to the control group (homozygous for major alleles at all three genetic loci) in an unpaired t-test. The study was terminated early because it was clear that we would not meet our recruitment targets and that the study was likely underpowered. Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — Probability that the observed difference was the result of random variation rather than a difference between the two populations; p = 0.92, t-test, 2 sided — No adjustment for multiple comparisons. Viewed as unnecessary inasmuch as none of the comparisons achieved p<0.05
Statistical Analysis 2: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.63, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 3: Comparison: Wild Type Genotype vs Missense Variant in SLC2A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.86, t-test, 2 sided — Not adjusted for multiple comparisons

2. Primary Outcome: Change in Fractional Excretion of Uric Acid (the Difference Between Data After Administration of Canagliflozin Minus Data Before Administration of Canagliflozin)
Description: For the study arm focused on individuals with a genetic variant in SLC2A9, the pharmacodynamic response to canagliflozin will be assessed by measuring the absolute change in fractional excretion of uric acid in the urine. Fractional excretion of uric acid represents the fraction of the calculated filtered uric acid load (serum uric acid level multiplied by the measured creatinine clearance rate) that was excreted in the urine.
Time Frame: 24 hour urine collection after administration of canagliflozin
Population: Data from all 30 patients are summarized. The primary statistical analysis is based on comparison of the 13 "wild type" genotype versus the 7 patients who are homozygous for the variant in SLC2A9 (GLUT9).
Measure: Mean (Standard Error); unit: absolute change in fractional excretion
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total Population
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
absolute change in fractional excretion | 0.25 (0.02) | 0.25 (0.02) | 0.28 (0.04) | 0.38 (0.05) | 0.29 (0.02)
Statistical Analysis 1: Comparison: Wild Type Genotype vs Missense Variant in SLC2A9; The study was terminated early because of slow recruitment. As a result the study did not achieve the statistical power that had been planned; Test type: Other — We compared the two groups ("wild type" versus SLC2A9 variant homozygotes. Null hypothesis: there are no differences between the two groups with respect to the pharmacodynamic effect of canagliflozin on fractional excretion of uric acid in the urine; p = 0.04, t-test, 2 sided — Because the study was terminated early, we did not have sufficient statistical power to adjust for multiple comparisons. We are reporting a nominal p-value without adjusting for multiple comparisons

3. Secondary Outcome: Canagliflozin-induced Change in Urinary Excretion of Sodium
Description: The pharmacodynamic response to canagliflozin will be assessed by measuring the % increase in 24 hour urinary excretion of sodium.
Time Frame: 24 hours after administration of canagliflozin
Measure: Mean (Standard Error); unit: % increase in urinary Na excretion
Groups:
- Total Population: Aggregate of all participants in the five study arms
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total Population
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
% increase in urinary Na excretion | 20 (12) | 66 (17) | 18 (10) | 48 (41) | 32 (11)
Statistical Analysis 1: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A4; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.07, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 2: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.53, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 3: Comparison: Wild Type Genotype vs Missense Variant in SLC2A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.92, t-test, 2 sided — Not corrected for multiple comparisons

4. Secondary Outcome: Canagliflozin-induced Change in Serum Creatinine
Description: The pharmacodynamic response to canagliflozin will be assessed by measuring changes in serum creatinine
Time Frame: 24 hours after administration of canagliflozin
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total Population
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
mg/dL | 0.06 (0.02) | -0.03 (0.02) | 0.07 (0.02) | 0.05 (0.02) | 0.04 (0.01)
Statistical Analysis 1: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A4; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.01, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 2: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.77, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 3: Comparison: Wild Type Genotype vs Missense Variant in SLC2A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.65, t-test, 2 sided — Not corrected for multiple comparisons

5. Secondary Outcome: Canagliflozin-induced Change in Serum Uric Acid
Description: The pharmacodynamic response to canagliflozin will be assessed by measuring changes in serum uric acid level
Time Frame: 24 hours after administration of canagliflozin
Population: Data from all 30 research participants will be summarized. Statistical analysis will focus on comparisons between the 13 participants who are homozygous for the major alleles at all three loci versus the three groups who are homozygous for each of the three other genetic variants.
Measure: Mean (Standard Error); unit: % change in serum uric acid level
Groups:
- Total Study Population: Aggregate of research participants in all four arms of the study
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total Study Population
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
% change in serum uric acid level | -22 (1.9) | -29 (4.2) | -12 (2.6) | -17 (3.0) | -20 (1.6)
Statistical Analysis 1: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A4; The "wild type" genotype group was compared to homozygotes for each of the three other genotypes; Test type: Other — Null hypothesis: None of the three genotypes is associated with an alteration in the pharmacodynamic effect of canagliflozin on urinary Na excretion; p = 0.20, t-test, 2 sided — Because the study was terminated early, the study does not have sufficient statistical power to adjust for multiple comparisons. Accordingly, nominal p-values are reported
Statistical Analysis 2: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Wild Type Genotype vs Missense Variant in SLC2A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.16, t-test, 2 sided — Not corrected for multiple comparisons

6. Secondary Outcome: Canagliflozin-induced Change in Fasting Plasma Glucose
Description: The magnitude of the change in fasting plasma glucose 24 hours after administration of canagliflozin (300 mg)
Time Frame: 24 hrs
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Wild Type Genotype | Nonsense Mutation in SLC5A4 | Nonsense Mutation in SLC5A9 | Missense Variant in SLC2A9 | Total Study Population
Number analyzed (Participants) | 13 | 4 | 6 | 7 | 30
mg/dL | -5.0 (1.5) | -2.0 (1.6) | -4.7 (2.8) | -3.4 (1.0) | -4.2 (0.9)
Statistical Analysis 1: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A4; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.21, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 2: Comparison: Wild Type Genotype vs Nonsense Mutation in SLC5A9; Null hypothesis: pharmacodynamic response is the same in the control group and homozygotes for the genetic variant; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.92, t-test, 2 sided — Not corrected for multiple comparisons
Statistical Analysis 3: Comparison: Wild Type Genotype vs Missense Variant in SLC2A9; Not corrected for multiple comparisons; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.39, t-test, 2 sided — Not corrected for multiple comparisons

ADVERSE EVENTS:
Time Frame: Participants received a single dose of canagliflozin (300 mg). The primary assessment of adverse events was during the 48 hours in which people were actively participating in the clinical trial (encompassing the two 24-hour urine collections).
Groups:
- Total Population of Participants in the Clinical Trial: All individuals received the same intervention. With such a small trial and so few adverse events, it is not meaningful to report adverse events for each arm separately. Adverse events were not collected or analyzed according to genotype status.
Arm/Group | Total Population of Participants in the Clinical Trial
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Population of Participants in the Clinical Trial (N=30)
Accident while driving a horse-drawn buggy (Musculoskeletal and connective tissue disorders) | 1 (1) — At a time when the participant was not taking the study drug (canagliflozin), the patient was driving a horse-drawn buggy and she experienced an accident without any significant injury.
Loose stools (Gastrointestinal disorders) | 1 (1) — One participant experienced loose stools within a few days of taking the single dose of canagliflozin (300 mg). It is unceratain whether this was related to the drug.

LIMITATIONS AND CAVEATS:
Small sample size: We had hoped to recruit more participants, but the need to collect two 24 hour urine samples turned out to be a major obstacle.

Small pilot study conducted in healthy volunteers rather than the target population for SGLT2 inhibitors.

Genetic studiy conducted in a Founder Population (Old Order Amish living in Lancaster County). Lancaster Amish chosen because of the availability of genotyping data and existence of infrastructure enabling genotype-directed "call-back" studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02462421/Prot_SAP_000.pdf